CLINICAL TRIAL: NCT03895736
Title: " Etude du Transcriptome Complet Lors du Syndrome Post-arrêt Cardiaque " Transcriptome Assessment After Cardiac Arrest
Brief Title: Transcriptome Assessment After Cardiac Arrest
Acronym: OMECARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other); University of Paris 5 - Rene Descartes (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Paris 12 Val de Marne University (Other); Ecole Nationale Vétérinaire d'Alfort (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00239-48; 2019-A00239-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-03-21; First posted 2019-03-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest After Initial Successful Resuscitation
Keywords: Transcriptome; messenger ribonucleic acid (mRNA); sequencing; biomarker; cardiac arrest; prognostication; successful resuscitation
MeSH Terms: conditions — Heart Arrest | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sampling — Sampling of 15 ml of blood during a blood test at Day 0, Day 1 and Day 3
  Other Names: Blood sampling at Day 0, Day 1 and Day 3

SUMMARY:
The purpose of this study is to determine whether the blood transcriptome of patients resuscitated after out-of-hospital could be an early predictor of the neurological outcome.

DETAILED DESCRIPTION:
Assessing the prognosis of the patients resuscitated after out-of-hospital cardiac arrest (OHCA) is still highly challenging. Beyond usual neurological markers, experimental and clinical studies have also shown that blood levels of several cytokines or miRNA could be significantly different after cardiac arrest in subjects prematurely died as compared to survivors with a good neurological recovery. Here the investigators propose to investigate a screening approach assessing simultaneously multiple targets of the post-cardiac arrest syndrome through analysis of the whole transcriptome of patients after OHCA. For this purpose, the investigators will collect blood samples from 60 patients after admission at hospital and then 1 and 3 days later. The Pittsburgh Cerebral Performance Category of each patient will be evaluated for each patient at day 60 after cardiac arrest. At the end of the collection period, the blood samples will be prepared for whole genome analysis and RNA sequencing. The primary analysis of the investigators will be the comparison of the transcriptome at day 0 after cardiac arrest in patients reaching Cerebral Performance Category (CPC) 1 at day 60 as compared to all other patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Delay between patients collapse and resumption of spontaneous circulation (ROSC) < 60 minutes
* Comatose patients ROSC with Glasgow score < 7
* Patient already registered in the social security system
* Consent of a family member, if able to understand in the emergency context, or attestation of emergency situation with a follow-up information notice

Exclusion Criteria:

* Cardiac arrest supposed to be provoked by trauma or sepsis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Early Transcriptome at hospital admission | Day 0
  Blood samples will be collected for each patient early after admission at hospital and blood whole transcriptome will be assessed by RNA sequencing
Pittsburgh Cerebral Performance Category at Day 60 | Day 60
  Pittsburgh Cerebral Performance Category will be evaluated for each patient at day 60

SECONDARY OUTCOMES:
Transcriptome at day 1 | Day 1
  Blood samples will be collected for each patient at day 1 and blood whole transcriptome will be assessed by RNA sequencing
Transcriptome at day 3 | Day 3
  Blood samples will be collected for each patient at day 3 and blood whole transcriptome will be assessed by RNA sequencing
Pittsburgh Cerebral Performance Category at Day 28 | day 28
  Pittsburgh Cerebral Performance Category will be evaluated for each patient at day 28
Number of participants with death at day 28 | day 28
Number of participants with death at day 60 | day 60

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cariou, Prof., Principal Investigator — Assistance Publique - Hôpitaux de Paris; Renaud Tissier, Prof, Study Chair — Ecole Nationale Vétérinaire d'Alfort
Locations (1):
- Hôpital Cochin, Assistance Publique Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No